CLINICAL TRIAL: NCT00088010
Title: Effects of Arzoxifene on Vertebral Fracture Incidence and on Invasive Breast Cancer Incidence in Postmenopausal Women With Osteoporosis or With Low Bone Density.
Brief Title: Effects of Arzoxifene on Bone Fractures and Incidence of Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8536; H4Z-MC-GJAD (Other: Eli Lilly and Company)
Record Dates: First submitted 2004-07-19; First posted 2004-07-20 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — LY 353381

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Arzoxifene
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Arzoxifene — 20mg, oral, tablet, once a day for 36 months
  Other Names: LY353381
  Arms: 1
Drug: Placebo — oral, tablet, once a day for 36 months
  Arms: 2

SUMMARY:
The purpose of this trial is to study:

* Effects of arzoxifene on bone fractures and bone mass.
* Effects of arzoxifene on getting breast cancer.
* Effects of arzoxifene on certain types of cardiovascular events, such as heart attack and stroke.
* Effects of arzoxifene that changes the amount of certain substances in the blood that are related to osteoporosis and cardiovascular health.
* Effects of arzoxifene on the uterus.
* The safety of arzoxifene and any side effects.

ELIGIBILITY:
Inclusion Criteria:

* 60-85 years of age
* Female
* At least two years since last menstrual cycle

Exclusion Criteria:

* Abnormal or unexplained vaginal bleeding.
* Bone disorders, other than osteoporosis or low bone mass
* History of breast cancer, cancer of the uterus, or any cancer in the last five years (except skin cancer).
* History of cerebral vascular accidents or venous thromboembolic events
* Medications outlined

Ages: 60 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9369 (Actual)
Dates: Start 2004-06; Primary Completion 2009-06 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Effects of arzoxifene on bone fractures and bone mass | 5 years
Effects of arzoxifene on getting breast cancer | 5 years
The safety of arzoxifene and any side effects | 5 years

SECONDARY OUTCOMES:
Effects of arzoxifene on certain types of cardiovascular events | 5 years
Effects of arzoxifene that changes the amount of certain substances in the blood that are related to osteoporosis and cardiovascular health | 5 years
Effects of arzoxifene on the uterus | 5 years
Effects of arzoxifene on cognition | 5 years
Effects of arzoxifene on back pain | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elk Grove, Illinois, United States

REFERENCES:
- [Derived] e Silva AV, Lacativa PG, Russo LA, de Gregorio LH, Pinheiro RA, Marinheiro LP. Association of back pain with hypovitaminosis D in postmenopausal women with low bone mass. BMC Musculoskelet Disord. 2013 Jun 12;14:184. doi: 10.1186/1471-2474-14-184. PMID 23758943
- [Derived] Powles TJ, Diem SJ, Fabian CJ, Neven P, Wickerham DL, Cox DA, Muram D, Agnusdei D, Dowsett SA, Amewou-Atisso M, Cummings SR. Breast cancer incidence in postmenopausal women with osteoporosis or low bone mass using arzoxifene. Breast Cancer Res Treat. 2012 Jul;134(1):299-306. doi: 10.1007/s10549-012-2041-5. Epub 2012 Apr 8. PMID 22484799
- [Derived] Goldstein SR, Bhattoa HP, Neven P, Cox DA, Dowsett SA, Alam J, Sipos A, Muram D. Gynecologic effects of arzoxifene in postmenopausal women with osteoporosis or low bone mass. Menopause. 2012 Jan;19(1):41-7. doi: 10.1097/gme.0b013e318223bbf4. PMID 21993078
- [Derived] Cummings SR, McClung M, Reginster JY, Cox D, Mitlak B, Stock J, Amewou-Atisso M, Powles T, Miller P, Zanchetta J, Christiansen C. Arzoxifene for prevention of fractures and invasive breast cancer in postmenopausal women. J Bone Miner Res. 2011 Feb;26(2):397-404. doi: 10.1002/jbmr.191. Epub 2010 Jul 23. PMID 20658564
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com